CLINICAL TRIAL: NCT04624009
Title: Relationship Between Near Infrared Spectroscopy Jugular Venous Oxygen Saturation (SjvO2) and Central Venous Saturation of Oxygen (ScvO2) in Critically Ill Patients.
Brief Title: Non-Invasive Measurement of SjvO2 Using Near Infrared Spectroscopy in Critically Ill Patients
Acronym: NIRS-SCJVO2
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Eduardo Schiffer, Professor, University Hospital, Geneva
Other Study IDs: SjvO2 vs ScvO2 / HUG-DMA
Record Dates: First submitted 2020-08-07; First posted 2020-11-10 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2022-05

CONDITIONS: Impaired Oxygen Delivery; Critically Ill Patient
Keywords: Brain oxygen delivery; Jugular Venous Oxygen Saturation; Central Venous Oxygen Saturation; Medical Device Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ScvO2 is an important parameter in the management of critically ill patient. The only way to measure it is to have an internal jugular or subclavian central venous catheter. With this trial, the investigators want to show a positive relationship between invasive ScvO2 measurement and noninvasive SjvO2 measurement with VO 100 medical device from Mespere LifeSciences, allowing the use of SjvO2 as a noninvasive surrogate of ScvO2 in critically ill patients.

DETAILED DESCRIPTION:
ScvO2 measures central venous oxygen saturation level from veins draining the head and upper body while SvO2 measures mixed venous oxygen saturation from the lower and upper half of the body. ScvO2 is more conveniently measured and less risky than Sv02 measurement although a central venous catheter is needed. ScvO2 gives knowledge about the balance between the delivery of oxygen and oxygen consumption in the body. Interest in ScvO2 monitoring in anesthesia and critical care has been debated. However, ScvO2 is still recommended as a major hemodynamic target of early resuscitation of critically ill patients. Even if ScvO2 measurement is far less invasive than SvO2 measurement through pulmonary artery catheter, it is accompanied with morbidity.

VO 100 medical device from Mespere LifeSciences allows a non-invasive measurement of SjvO2 using the NIRS technique. Jugular venous oxygen saturation (SjvO2) is a measurement of the amount of oxygen left in the venous system after the brain has removed the oxygen that it needs.

On the same principle that a positive relationship between ScvO2 and SvO2 has been shown, what the investigators are trying to do is to show a positive relationship between SjvO2 and ScvO2 in order to possibly use in the future SjvO2 measured by VO 100 as a noninvasive surrogate of ScvO2.

ELIGIBILITY:
Inclusion Criteria:

* all ICU adult patients routinely equipped with a central venous catheter placed in internal jugular or subclavian vein allowing ScvO2 measurement from blood sampling.

The investigators will perform this study only on patients already equipped with an internal jugular CVC. In other words, the placement of the CVC is not conditioned by the study realization.

Exclusion Criteria:

* patients with CVC placed in another site than internal jugular vein.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ICU adult patients routinely equipped with a central venous catheter placed in internal jugular or subclavian vein
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Comparison of venous oxygen saturation 1 | On admission to the intensive care unit
  Comparison of ScvO2 values from CVC blood sample and SjvO2 values from the VO 100 (% oxygen saturation)

SECONDARY OUTCOMES:
Comparison of venous oxygen saturation 2 | 3 days after admission into the intensive care unit
  Comparison of ScvO2 values from CVC blood sample and SjvO2 values from the VO 100 (% oxygen saturation)
Comparison of venous oxygen saturation 3 | On admission to internal medicine ward
  Comparison of ScvO2 values from CVC blood sample and SjvO2 values from the VO 100 (% oxygen saturation)

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - University of Geneva, Geneva
  - Eduardo Schiffer, Veyrier